CLINICAL TRIAL: NCT00109928
Title: Phase II Trial of Cisplatin Plus Etoposide Plus Gemcitabine Plus Solumedrol (PEGS) in Peripheral T-Cell Non-Hodgkin's Lymphoma
Brief Title: S0350 Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage II, Stage III, or Stage IV Peripheral T-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000425643; S0350 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Lymphoma
Keywords: stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic | interventions — Cisplatin; Etoposide; Gemcitabine; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEGS Treatment (Experimental): VP-16 (Etoposide) 40 mg/m2 IV Days 1-4 Methyl Prednisolone 250 mg IV Days 1-4 Cisplatin 25 mg/m2 IV Days 1-4 Gemcitabine 1,000 mg/m2 IV Day 1
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: gemcitabine; Drug: methylprednisolone

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Drug: gemcitabine
Drug: methylprednisolone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, etoposide, gemcitabine, and methylprednisolone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating patients with newly diagnosed stage II, stage III, or stage IV T-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine 2-year overall survival of patients with newly diagnosed, bulky stage II or stage III or IV peripheral T-cell non-Hodgkin's lymphoma treated with cisplatin, etoposide, gemcitabine, and methylprednisolone.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the response rate (complete unconfirmed response, complete response, and partial response) in patients treated with this regimen.
* Determine progression-free survival of patients treated with this regimen.

OUTLINE: This is a pilot, multicenter study.

Patients receive cisplatin IV over 30-60 minutes, etoposide IV over 30-60 minutes, and methylprednisolone IV over 5 minutes on days 1-4. Patients also receive gemcitabine IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 3-6 weeks, 3 months, and then every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of peripheral T-cell non-Hodgkin's lymphoma

  * Newly diagnosed, relapsed or progressing disease after 1 prior treatment with a non-platinum based chemotherapy (e.g., CHOP)
  * Bulky stage II or stage III or IV disease
* The following histologies are not eligible:

  * T-cell prolymphocytic leukemia
  * T-cell large granular lymphocytic leukemia
  * Any NK-cell leukemia
  * Adult T-cell leukemia/lymphoma
  * Mycosis fungoides/Sézary syndrome
  * Lymphomatoid papulosis
  * Nasal-type extranodal NK/T-cell lymphoma
  * Enteropathy-type T-cell lymphoma
  * Hepatosplenic T-cell lymphoma
  * Subcutaneous panniculitis-like T-cell lymphoma
  * Angioimmunoblastic T-cell lymphoma
  * Primary cutaneous anaplastic large cell lymphoma (ALCL)
  * ALCL with CD30, ALK, and EMA expression

    * ALCL morphology that fails to express ALK or EMA allowed provided T-cell lineage is confirmed by immunotyping or genetic testing
* Bidimensionally measurable disease
* Adequate samples (e.g., core biopsies, especially multiple core biopsies) from the original diagnostic specimen available

  * Needle aspiration or cytology is not considered adequate samples
* No clinical evidence of Central nervous system (CNS) involvement by lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2 times upper limit of normal

Renal

* Creatinine clearance ≥ 30 mL/min

Cardiovascular

* No history of congestive heart failure
* No history of myocardial infarction
* No history of unstable angina
* No history of asymptomatic arrhythmias
* Ejection fraction normal by multigated acquisition (MUGA) scan (for patients with questionable cardiac history)
* No other history of impaired cardiac status

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* Mild clinical hearing loss allowed provided patient is willing to accept the potential for worsening of hearing loss
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Must have had a chest x-ray or CT scan of the chest and a CT scan of the abdomen and pelvis within the past 28 days

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior biologic therapy
* No concurrent routine use of bone marrow colony-stimulating factors

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for this cancer
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No prior cytotoxic therapy for this cancer
* Concurrent enrollment in SWOG-8819 or SWOG-8947 allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-09; Primary Completion 2012-06 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daruka Mahadevan, MD, PhD, Study Chair — University of Arizona
Locations (77):
- United States (77):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Mahadevan D, Unger JM, Spier CM, Persky DO, Young F, LeBlanc M, Fisher RI, Miller TP. Phase 2 trial of combined cisplatin, etoposide, gemcitabine, and methylprednisolone (PEGS) in peripheral T-cell non-Hodgkin lymphoma: Southwest Oncology Group Study S0350. Cancer. 2013 Jan 15;119(2):371-9. doi: 10.1002/cncr.27733. Epub 2012 Jul 25. PMID 22833464

RESULTS

PARTICIPANT FLOW:
Groups:
- PEGS: Patients received IV cisplatin 25 mg/m2 days 1-4, etoposide 40 mg/m2 days 1-4, gemcitabine 1000 mg/m2 day 1 and solumedrol 250 mg days 1-4 of a 21 day cycle for 6 cycles.
Period: Overall Study
Arm/Group | PEGS
Started | 34
Eligible | 33
Eligible and Began Protocol Therapy | 33
Completed | 21
Not Completed | 13
Not completed — Adverse Event | 2
Not completed — Progression | 6
Not completed — Death | 2
Not completed — not protocol specified | 2
Not completed — not eligible | 1

BASELINE CHARACTERISTICS:
Population: Peripheral T-cell lymphomas (PTCLs) with stage II bulky, III or IV with extra-nodal, nodal and transformed cutaneous presentations were eligible.
Arm/Group | PEGS
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 60 [20 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 2-year Overall Survival Rate
Description: The overall survival rate is the percentage of patients who are alive 2 years after registration to the study. Overall survival is defined as the time between study registration and death due to any cause.
Time Frame: 0-2 years
Population: All eligible patients who started protocol treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEGS
Number analyzed (Participants) | 33
percentage of participants | 31 [8 to 54]

2. Secondary Outcome: 2-year Progression-free Survival Rate
Description: Progression-free survival rate is the percentage of patients who do not show signs of progression at 2 years after registration to the study, including those whose disease has either completely or partially responded to treatment, or those whose disease is stable. Progression-free survival is defined as the time between study registration and documented progression, or death if no progression was observed.
Time Frame: 0-2 years
Population: All eligible patients who started protocol treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEGS
Number analyzed (Participants) | 33
percentage of participants | 12 [0.1 to 31]

3. Secondary Outcome: Response Rate
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: up to 3 years or time of disease progression
Population: All eligible patients who started protocol treatment were included in the analysis.
Measure: Number; unit: participants
Arm/Group | PEGS
Number analyzed (Participants) | 33
participants
  Complete Response | 6
  Unconfirmed Complete Response | 2
  Partial Response | 5
  No Response | 20

4. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: up to 18 weeks of protocol treatment
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- PEGS: Patients received IV cisplatin 25 mg/m2 days 1 to 4, etoposide 40 mg/m2 days 1 to 4, gemcitabine 1000 mg/m2 day 1 and solumedrol 250 mg days 1 to 4 of a 21 day cycle for 6 cycles.)
Arm/Group | PEGS
Number analyzed (Participants) | 33
Participants
  Albumin, serum-low (hypoalbuminemia) | 1
  Allergic reaction/hypersensitivity | 1
  Anorexia | 2
  Ataxia (incoordination) | 1
  Auditory/Ear-Other (Specify) | 1
  Blood/Bone Marrow-Other (Specify) | 1
  Colitis, infectious (e.g., Clostridium difficile) | 2
  Creatinine | 2
  Diarrhea | 2
  Dysphagia (difficulty swallowing) | 1
  Dyspnea (shortness of breath) | 1
  Fatigue (asthenia, lethargy, malaise) | 2
  Febrile neutropenia | 4
  Gastrointestinal-Other (Specify) | 1
  Glucose, serum-high (hyperglycemia) | 4
  Glucose, serum-low (hypoglycemia) | 1
  Hemoglobin | 9
  Hemorrhage, CNS | 1
  Hypotension | 2
  Incontinence, anal | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Bladder | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1
  Leukocytes (total WBC) | 8
  Lymphopenia | 7
  Magnesium, serum-low (hypomagnesemia) | 2
  Nausea | 1
  Neurology-Other (Specify) | 1
  Neuropathy: motor | 1
  Neuropathy: sensory | 2
  Neutrophils/granulocytes (ANC/AGC) | 16
  Pain - Abdomen NOS | 1
  Platelets | 8
  Potassium, serum-low (hypokalemia) | 1
  Renal failure | 2
  Sodium, serum-low (hyponatremia) | 2
  Thrombotic microangiopathy | 1
  Tinnitus | 1
  Tumor lysis syndrome | 1
  Uric acid, serum-high (hyperuricemia) | 1

ADVERSE EVENTS:
Time Frame: up to 18 weeks of protocol treatment
Groups:
- PEGS: Patients received IV cisplatin 25 mg/m2 days 1-4, etoposide 40 mg/m2 days 1-4, gemcitabine 1000 mg/m2 day 1 and solumedrol 250 mg days 1-4 of a 21 day cycle for 6 cycles.)
Arm/Group | PEGS
Serious Adverse Events (participants affected / at risk) | 5/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEGS (N=33)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemorrhage, CNS (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEGS (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 28
Cardiac General-Other (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 2
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 2
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 3
Auditory/Ear-Other (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 5
Ocular/Visual-Other (Eye disorders) | 2
Ascites (non-malignant) (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 14
Distention/bloating, abdominal (Gastrointestinal disorders) | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 24
Pain - Abdomen NOS (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 11
Edema: head and neck (General disorders) | 2
Edema: limb (General disorders) | 16
Edema: trunk/genital (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 6
Injection site reaction/extravasation changes (General disorders) | 2
Pain - Chest/thorax NOS (General disorders) | 2
Pain-Other (General disorders) | 9
Rigors/chills (General disorders) | 6
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Oral cav (Infections and infestations) | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 3
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4
AST, SGOT (Investigations) | 7
Alkaline phosphatase (Investigations) | 7
Bilirubin (hyperbilirubinemia) (Investigations) | 3
Creatinine (Investigations) | 15
INR (of prothrombin time) (Investigations) | 2
Leukocytes (total WBC) (Investigations) | 20
Lymphopenia (Investigations) | 11
Metabolic/Laboratory-Other (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 21
Platelets (Investigations) | 18
Weight gain (Investigations) | 8
Weight loss (Investigations) | 4
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 10
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 15
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 9
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 6
Pain - Back (Musculoskeletal and connective tissue disorders) | 6
Pain - Bone (Musculoskeletal and connective tissue disorders) | 4
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 4
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2
Pain - Neck (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 6
Neurology-Other (Nervous system disorders) | 4
Neuropathy: sensory (Nervous system disorders) | 11
Ocular/Visual-Other (Nervous system disorders) | 2
Pain - Head/headache (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 2
Taste alteration (dysgeusia) (Nervous system disorders) | 5
Confusion (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 9
Mood alteration - agitation (Psychiatric disorders) | 2
Mood alteration - anxiety (Psychiatric disorders) | 9
Mood alteration - depression (Psychiatric disorders) | 2
Glomerular filtration rate (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 12
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 2
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 3
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 15
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No